CLINICAL TRIAL: NCT02279979
Title: Thoratec Corporation HeartMate PHP™ Cardiogenic Shock Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thoratec HeartMate PHP™ CS
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Cardiogenic Shock
Keywords: PHP; Cardiogenic Shock; Percutaneous; Ventricular Assist; Heart Pump; Catheter; Thoratec Corporation
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): All enrolled patients will be treated with the HeartMate PHP device
  Interventions: Device: HeartMate PHP

INTERVENTIONS:
Device: HeartMate PHP — The HeartMate PHP system is a catheter-based heart pump and console designed to provide hemodynamic left ventricular support for up to 3 days to stabilize patients by maintaining adequate systemic cardiac output.

SUMMARY:
The primary objective of this study is to assess reasonable safety and performance of the HeartMate PHP to provide hemodynamic support for up to 72 hours in patients with cardiogenic shock requiring stabilization.

DETAILED DESCRIPTION:
The HeartMate PHP is a catheter-based axial flow pump designed to provide partial left ventricular circulatory support. This prospective, nonrandomized, controlled, single-arm, multi-center, open-label trial will evaluate the safety and performance of the device in patients with cardiogenic shock.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is indicated for left ventricular support according to current medical guidelines ("current medical guidelines" applies only to patients enrolled in Germany)
2. Patient has a cardiac index of < 2.2 L/min/m2 and is being treated with at least one moderate dose inotrope or at least one moderate dose of vasopressor (e.g., milrinone ≥0.3 mcg/kg/min, dopamine > 5 mcg/kg/min, dobutamine > 5 mcg/kg/min) AND:

   * PCWP > 18 mmHg, AND
   * Systolic blood pressure < 100 mmHg, AND
   * Decreased organ perfusion as evidenced by urine output of 50 mL/hr OR increased creatinine of 0.3 mg/dl from baseline obtained within 2 weeks, OR cool extremities
3. Written, signed, and dated informed consent

Exclusion Criteria:

1. Patient is >85 years of age
2. Right ventricular failure requiring mechanical circulatory support
3. ST elevation myocardial infarction (STEMI) within 30 days of procedure
4. Cardiac arrest within 7 days of procedure requiring CPR
5. Current treatment with mechanical circulatory device such as IABP, ECMO, centrifugal pump, etc.
6. Documented acute myocarditis
7. Active major cardiac rhythm disturbances (e.g., ventricular tachycardia, ventricular fibrillation).
8. Hypertrophic disease or any left ventricular outflow tract obstruction
9. Active sepsis defined as bacteremia, fever ≥ 101.5 degrees F
10. Mural thrombus in the left ventricle
11. History of aortic valve replacement
12. End-stage renal disease requiring dialysis
13. Documented presence of aortic stenosis (orifice area of 1.5 cm2 or less)
14. Moderate to severe aortic insufficiency (echocardiographic assessment of aortic insufficiency graded as 2 or higher)
15. Platelet count < 100,000
16. Allergy or Intolerance to heparin, aspirin, clopidogrel, ionic and nonionic contrast media, or any other potentially required anticoagulants or antiplatelet therapy drugs
17. Known coagulopathies
18. Presence of risk factors for severe liver and/or renal dysfunction
19. Stroke within 90 days of enrollment
20. Significant peripheral vascular disease
21. History of heparin induced thrombocytopenia
22. Patient is pregnant or planning to become pregnant during the study period
23. Patient is breastfeeding.
24. Any active disease (e.g., active cancer) which could affect the patient's participation in the study, or if life expectancy is less than 1 year.
25. Any active disease in which the investigator determines would make the patient an inappropriate candidate for the study.
26. Participation in another clinical study of an investigational drug or device that has not met its primary endpoint

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Clinical stabilization defined as improvement of Cardiac Index to > 2.2 L/min/m2 | 72 hours

SECONDARY OUTCOMES:
An assessment of major adverse events | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Chatterjee, Study Director — Thoratec LLC, St. Jude Medical, Abbott
Locations (6):
- Czechia (2):
  - Na Homolce Hospital, Prague
  - Institute for Clinical and Experimental Medicine (IKEM), Prague
- Germany (2):
  - Universitätskliniken Düsseldorf, Düsseldorf
  - Medizinische Hochschule Hannover, Hanover
- Semmelweis University Heart and Vascular Center, Budapest, Hungary
- Erasmus Medical Center, Rotterdam, Netherlands